CLINICAL TRIAL: NCT02871362
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Benefit of IQP-AS-118 on Blood Pressure and LDL-cholesterol: A Pilot Study
Brief Title: Benefit of IQP-AS-118 on Blood Pressure and LDL-cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INQ/030915
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Blood Pressure; Low Density Lipoprotein Cholesterol Level

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IQP-AS-118 (Experimental): To be taken once daily with a glass of water. The tablets should not be chewed, but swallowed whole.
  Interventions: Dietary Supplement: IQP-AS-118
- Placebo (Placebo Comparator): To be taken once daily with a glass of water. The tablets should not be chewed, but swallowed whole.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IQP-AS-118 — Take one a day
  Arms: IQP-AS-118
Dietary Supplement: Placebo — Take one a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the benefit and tolerability of IQP-AS-118 on the systolic and diastolic blood pressure (BP) and to explore the effects on parameters of lipid metabolism in subjects with elevated BP and low density lipoprotein cholesterol (LDL-C) levels in a pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian males and females, 18-65 years of age
2. Body mass index (BMI) 18.5-29.9 kg/m2
3. Generally in good health, in particular an electrocardiogram (ECG) without pathological findings at screening
4. High normal BP levels (130-139 / 85-89) for 20% of randomized subjects and hypertension grade 1 (140-159 / 90-99) BP levels for 80% of randomized subjects at screening (mean of the 2nd and 3rd measurement during the assessment in triplicate at screening) and at baseline (mean of the 2nd and 3rd measurement during the assessment in triplicate at week 0)
5. LDL-C 100-159 mg/dL
6. Readiness to comply with study procedures, in particular:

   * Consumption of the IP during the entire study
   * Maintaining the habitual diet, with the exception of consumption of maximal 2 garlic cloves per week
   * Accepting blood draws
   * Complying with requirements for BP measurements (such as avoiding any strenuous exercise and stimulants (alcohol, caffeine) for at least 24 h before the measurement; refraining from extreme cold and heat exposure and food and fluid intake for at least 1 h before the measurement)
   * Filling in health questionnaires
7. Non-smoker / smoking cessation of last ≥12 months prior to screening
8. Stable body weight in the last 3 months prior to screening (<3 kg self-reported change)
9. If allowed concomitant medications are taken this must have been stable at least during the last month prior to screening
10. Women of child-bearing potential only:

    1. negative pregnancy testing (ß-HCG in urine at screening)
    2. commitment to use reliable contraception methods during the entire study Participation is based upon written informed consent form (ICF) by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Known sensitivity to any components of the IP
2. Clinically significant disturbances in lipid metabolism
3. Known genetic hyperlipidemia
4. Known secondary hypertension
5. Known white-coat hypertension
6. Known type-1-diabetes
7. Uncontrolled or within the last 6 months prior to screening diagnosed type-2-diabetes
8. Untreated or non-stabilized thyroid disorder
9. History and/or presence of clinically significant cardiovascular disease as per investigator's judgement:

   1. Known congenital heart defects
   2. Myocardial infarction, heart failure, angina pectoris, life-threatening arrhythmia or stroke within the last 6 months prior to screening
   3. Existing thrombosis or disposition to thrombosis
10. Any other known significant or serious condition / disease that renders subjects ineligible, e.g.:

    1. History of malignancy within the past 5 years prior to screening
    2. Bleeding disorder and/or need for anticoagulants (anti-platelet agents are allowed)
    3. Current psychiatric care and/or use of neuroleptics
    4. Bariatric surgery in the last 12 months prior to screening
11. Any known metabolic disease, gastrointestinal disorder or other clinically significant disease/disorder which in the investigator's opinion could interfere with the results of the study or the safety of the subject
12. Known arm lymphedema (e.g. due to mastectomy)
13. Other clinically relevant excursions of safety parameters and/or deviations > 2 x ULN (upper limit of normal)
14. Dietary habits that may interfere with the study objectives:

    1. Eating disorder
    2. Subjects with dietary restriction that may affect the study outcome
    3. Participation in a weight loss program
15. Use of drugs or supplements that can influence SBP or DBP (e.g. ACE inhibitors, diuretics, calcium channel or ß-blockers, grape seed extract, coenzyme Q10 etc.) within the last 4 weeks prior to screening and during the study
16. Use of lipid lowering drugs (affecting lipid metabolism, platelet function or antioxidant status, etc.) OR dietary or health supplements (e.g. omega-3 fatty acids, green tea extract, calcium, red yeast rice, phytosterols (incl. enriched products such as e.g. Becel), oat fiber, niacin, soy protein, psyllium seed husk, glucomannan, chitosan or probiotics/prebiotics) within the last 4 weeks prior to screening and during the study
17. Use of drugs that can influence cholesterol levels (e.g. corticosteroids, amiodarone, estrogen, anabolic ster-oids)
18. Use of weight loss treatment
19. Use of any recreational drugs
20. Alcohol abuse (men: ≥21 units/week, women: ≥14 units/ week; 1 unit equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
21. Women of child-bearing potential: pregnant or breast-feeding
22. Participation in another study or blood donation during the last 30 days prior to screening
23. Any other reason deemed suitable for exclusion as per investigator's judgment, e.g.:

    1. Insufficient compliance with study procedures
    2. Inability to communicate with the site study staff

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure (Systolic & Diastolic) | 12 weeks
  Week 12 vs. week 0

SECONDARY OUTCOMES:
Systolic blood pressure | 12 weeks
  Week 4 and week 8 vs. week 0, respectively
Diastolic blood pressure | 12 weeks
  Week 4 and week 8 vs. week 0, respectively
Fasting LDL-C concentration and non-HDL-C | 12 weeks
  Week 12 vs. week 0
Fasting TC Concentration | 12 weeks
  Week 12 vs. week 0
Fasting HDL-C Concentration | 12 weeks
  Week 12 vs. week 0
Fasting TG Concentration | 12 weeks
  Week 12 vs. week 0
Fasting LDL-C/HDL-C and TC/HDL-C ratio | 12 weeks
  Week 12 vs. week 0
Fasting Lp (a) concentrations | 12 weeks
  Week 12 vs. week 0
hs-CRP | 12 weeks
  Week 12 vs. Screening
Homocysteine | 12 weeks
  Week 12 vs. Screening
Pulse wave assessment | 12 weeks
  Week 12 vs. week 0
Metabolome analysis | 12 weeks
  Week 12 vs. week 0
SF-12 | 12 weeks
  Week 4, week 9 and week 12 vs. week 0, respectively
Global evaluation of benefit by the subjects/ investigator | 12 weeks
  Week 12 only

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, MD, phD, Principal Investigator — analyze & realize GmbH
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No